CLINICAL TRIAL: NCT04373278
Title: Infection After Free Fibula Flap Reconstruction of the Mandible: a Retrospective Cohort Study
Acronym: FibFlapI
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Principal Investigator, Eugénie MABRUT, clinical research asssistant, Hospices Civils de Lyon
Other Study IDs: 19-273
Record Dates: First submitted 2020-04-30; First posted 2020-05-04 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Bone and Joint Infection
Keywords: mandibular; flap

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- description of infection of free fibula flap reconstruction
  Interventions: Other: failure of reconstruction of the mandibule by free fibula flap

INTERVENTIONS:
Other: failure of reconstruction of the mandibule by free fibula flap — description of failure of reconstruction of the mandibule by free fibula flap:delay, type of bacteria involved in the failure, treatment, outcome

SUMMARY:
Mandibular osteitis after flap reconstruction is rare but is a serious infection with significant sequelae.

The aim of this study is to describe this type of infection

ELIGIBILITY:
Inclusion Criteria:

* patients having had infection after a free bony flap reconstruction of the mandibule treated as an osteomyelitis at the CRIOAc between 2014 and 2020

Exclusion Criteria:

* non-bony flap

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients having had infection after a free flap reconstruction of the mandibule
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
rate of failure after free fibula flap reconstruction of the mandible | Outcome is measured at the end of follow-up (usually between 12 and 24 months after antibiotic therapy disruption]
  description of failure after free fibula flap reconstruction of

SECONDARY OUTCOMES:
rate of bacteria involved in failure after free fibula flap reconstruction of the mandible | when bacteria had growth up on culture; usually 2-3 weeks after the sample extracted on the surgery
  epidemiology of bacteria which causes the failure

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://www.crioac-lyon.fr